CLINICAL TRIAL: NCT01032226
Title: Evaluation of CNAP During Induction and Maintenance of General Anesthesia
Brief Title: Evaluation of CNAP During Anesthesia
Acronym: CnapEval
Status: Terminated | Type: Observational
Why Stopped: Difficulty to include more patients
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/03
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: General Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare

* the non invasive measurement of arterial pressure (CNAP monitor)
* with the invasive measurement of arterial pressure (radial artery catheter) during induction and maintenance of general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* ASA II, III or IV
* weight between 40 and 180 kg; BMI < 35
* surgical procedure performed in supine position
* normal Allen's test and hand Doppler examination.

Exclusion Criteria:

* cardiac arrhythmias,
* history of vascular surgery or vascular implant in the upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major surgery with the need for an invasive blood pressure measurement
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Comparison between both methods of arterial pressure measurement | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France